CLINICAL TRIAL: NCT03520660
Title: Long-Term Follow-Up Of Subjects With CHC Who Achieved A Sustained Virological Response Following Therapy With Direct Acting Antiviral Agents
Brief Title: People With CHC Who Achieved a Sustained Virological Response Following Therapy With Direct Acting Antiviral Agents
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180091; 18-DK-0091
Record Dates: First submitted 2018-05-09; First posted 2018-05-11 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01-09

CONDITIONS: Diabetes Mellitus; Hepatitis C, Chronic; Cardiovascular Diseases
Keywords: Natural History; Hepatitis C Virus; Hepatocellular Carcinoma; Fibrosis; Immune Response
MeSH Terms: conditions — Diabetes Mellitus; Hepatitis C, Chronic; Cardiovascular Diseases; Hepatitis C; Carcinoma, Hepatocellular; Fibrosis | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase I (Experimental): Phase I treatment
  Interventions: Drug: Epclusa
- Phase II after Phase I (No Intervention): Participants who achieved SVR12 in Phase I
- Phase II without Phase I (No Intervention): Participants who achieved SVR 24 previously

INTERVENTIONS:
Drug: Epclusa — sofosbuvir/velapatasvir combination (Epclusa)
  Arms: Phase I

SUMMARY:
Background:

Chronic hepatitis C infects the liver. It may scar the liver. This is called cirrhosis and may lead to liver cancer or death. Current chronic hepatitis C treatments cure most people. But some keep getting complications even after it is cured. Researchers want to study why.

Objective:

To study the course and complications of liver disease after cure of hepatitis C infection.

Eligibility:

Adults 18 years and older infected with chronic hepatitis C virus who were never treated or were treated and not cured and those who were cured

Design:

Participants will be screened with:

Blood and urine tests

Questionnaires

Liver ultrasound

Fibroscan. A probe vibrates the liver, testing stiffness.

In Phase 1, people with chronic hepatitis C will:

Have a 3-day hospital admission to repeat some screening tests and have a liver biopsy. A small piece of liver is removed by needle passed through the skin.

Take 1 tablet containing 2 hepatitis C drugs once a day for 12 weeks.

Repeat some blood tests at 3 visits in those 12 weeks while on treatment, then 4 additional visits in the next 24 weeks with more blood work collected.

Phase 1 participants who test negative for hepatitis C and all other eligible participants will enter Phase 2.

Phase 2 participants will have a visit every 24 weeks for 10 years. These may include:

Repeats of screening tests

Questionnaires

Scans

Stool tests

Chest x-ray

Heart function test

Endoscopy. A tube guides a camera into the upper digestive system.

At about 5 years, participants will have another liver biopsy.

Some participants will give separate consent for genetic testing and a special blood procedure.

DETAILED DESCRIPTION:
Study Description:<TAB>

We intend to enroll up to 350 subjects with chronic hepatitis C virus (HCV) infection. Subjects will be recruited from two sources:

1. Phase I: treatment na(SqrRoot) ve or experienced who have failed a prior treatment (including DAA-experienced) who are willing to undergo a pre-treatment liver biopsy.

   1. Subjects yet to achieve an SVR will receive 12 weeks of therapy with sofosbuvir/velapatasvir (Epclusa(R)) fixed dose combination
   2. Subjects yet to achieve SVR with evidence of clinical cirrhosis will undergo a transjugular liver biopsy with hepatic venous portal gradient (HVPG) pressure measurements in lieu of the percutaneous liver biopsy
2. Phase II: subjects who have already achieved sustained virologic response (SVR) with oral direct-acting antiviral agent (DAA) only regimen and who have undergone a liver biopsy prior to therapy and no history of hepatic decompensation or hepatocellular carcinoma.

   Subjects who have attained an SVR prior to enrollment (or upon achieving an SVR12 and SVR24 in Phase I) will undergo a thorough medical evaluation:
   * laboratory testing
   * Fibroscan(R)
   * hepatic ultrasound

   Thereafter, subjects will be followed prospectively every 24 weeks for liver decompensation (ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, variceal hemorrhage), hepatocellular carcinoma, liver-related mortality, and all-cause mortality. During each study visit, subjects will be questioned on the development of these adverse outcomes. In addition, blood will be drawn for the assessment of routine blood tests, quantitative viral biomarker levels, serological response markers and immune cell functional status. Blood, urine, and stool will be collected and stored for exploratory biomarker development. Fibroscan(R) will be performed annually in all subjects. For subjects with cirrhosis, esophagogastroduodenoscopy (EGD) will be performed annually and imaging every 24 weeks. At the end of 240 weeks, all subjects will be admitted for a liver biopsy to assess the stage of liver fibrosis. In subjects with cirrhosis at study entry, the liver biopsy will be performed by the transjugular route with hepatic venous portal gradient (HVPG) pressure measurements.

   The primary goal of the study will be to describe the outcome of viral eradication following treatment with direct acting antiviral agents, to identify predictors of adverse outcomes after sustained viral eradication and regression of fibrosis/cirrhosis.

   Objectives:

   Primary Objective:
   * Phase 1: SVR12 and SVR24
   * Phase II: The rate of clinical outcomes (ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, variceal hemorrhage), hepatocellular carcinoma, liver-related mortality, and all-cause mortality

   Secondary Objectives:
   * Phase II: The proportion and rates of fibrosis regression in subjects
   * Phase II: The agreement between Fibroscan and Ishak fibrosis score
   * Phase II: The comparison of change in Fibroscan and change in Ishak fibrosis as predictors of the primary outcome.
   * Phase II: To assess regression of portal hypertension in subjects with pre-existing portal hypertension either confirmed by direct portal pressure measurement, indirectly by hepatic venous pressure gradient or clinical evidence of portal hypertension such as presence of esophageal or gastric varices of portal hypertensive gastropathy and all-cause mortality.

   Exploratory Objective:
   * To develop novel biomarkers and genetic predictors of liver-related complications including hepatocellular carcinoma.
   * To assess outcome of HCV-related immune dysfunction following sustained eradication of HCV.
   * To assess changes in antibody titer and breadth, B cell activation, and T cell memory after sustained HCV eradication.
   * To prospectively assess the rate of non-hepatic outcomes (diabetes, cardiovascular and renal disease, malignancy including lymphoma, and health related quality of life) following SVR with DAA agents.
   * To characterize the changes in serum lipids and lipoproteins during and after therapy with direct acting antiviral agents and assess cardiovascular risk following eradication of HCV based on serum/plasma LDL particle number.

   Endpoints:

   Primary Endpoint:
   * SVR at 12 weeks after completion of 12 weeks of treatment.
   * Composite of ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, variceal hemorrhage, hepatocellular carcinoma, liver-related mortality, and all-cause mortality at 480 weeks.

   Secondary Endpoints:
   * Improvement in semi-quantitative Ishak fibrosis score after HCV clearance.
   * Correlation between Fibroscan (transient elastography) with Ishak fibrosis score after HCV clearance.
   * Does change improvement in Fibroscan and change in Ishak fibrosis correlate with clinical outcome.
   * Change in portal pressure after SVR12.

ELIGIBILITY:
* INCLUSION CRITERIA:

Phase I Treatment

* Male or female >= 18 years of age
* Either treatment naive or experienced defined as failure of a prior course of interferon-based and ribavirin, DAA plus interferon and DAA only
* Confirmation of chronic HCV infection documented by:

  * A positive HCV RNA or positive HCV genotyping test at least 6-months prior to the Baseline/Day 1 visit
  * A liver biopsy performed prior to screening visit showing evidence of chronic hepatitis.
* Subjects must have the following laboratory parameters at screening:

  * ALT <= 10 x the upper limit of normal (ULN)
  * AST <= 10 x ULN
  * Total bilirubin <2.5 mg/dL, Direct bilirubin <= 1.5 ULN
  * Platelets >= 50,000 K/mm^3
  * HbA1c <= 8.5%
  * Hemoglobin >= 10g/dL
  * Albumin >= 3g/dL
  * INR <= 1.5 unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR.
  * HCV RNA positive at screening.
* Subjects must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator.

Phase II Follow-up

* Male or female >= 18 years of age.
* SVR24 following therapy with a direct acting antiviral agent regimen and available liver biopsy performed prior to treatment.
* Subject must be of generally good health as determined by the Investigator.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

Phase I Treatment

* Pregnancy or lactation
* Inability to practice one form of adequate contraction for females of childbearing potential
* Prior treatment with a NS5a agent
* Current or prior history of any of the following:

  * Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol; subjects currently under evaluation for a potentially clinically significant illness (other than HCV) are also excluded
  * Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug
  * Decompensated liver disease as defined by serum bilirubin >= 2.5 mg/dL (with direct bilirubin >= 1.5 mg/dL), INR >1.5 a serum albumin of less than 3 g/dL, or a history of ascites, hepatorenal syndrome, variceal bleeding, or hepatic encephalopathy
  * Solid organ transplantation
  * Significant pulmonary disease, significant cardiac disease
* History of malignancy or treatment for a malignancy within the past 3 years that is associated with a life expectancy <5 years (except adequately treated carcinoma in situ or basal cell carcinoma of the skin).
* Chronic liver disease of a non-HCV etiology with the exception of steatosis (e.g., chronic hepatitis B, hemochromatosis, Wilson s disease, alfa-1 antitrypsin deficiency, cholangitis).
* Evidence of harmful or hazardous drinking as defined as a score >= 8 on the AUDIT questionnaire.
* Co-infection with HIV defined as the presence of anti-HIV in serum.
* Clinically relevant drug abuse based on patient history within 12 months of screening.
* Use of medications contraindicated with use of sofosbuvir/velpatasvir within 21 days of the Baseline/Day 1 visit; this washout period does not apply to proton pump inhibitors, which can be taken up to 7 days before baseline Day 1 for the following:

  * Acid reducing Agents
  * Antiarrhythmics
  * Anticancer
  * Antimycobacterial
  * HIV antivirals
  * Herbal supplements
  * HMG-CoA Reductase Inhibitors
* Use of antiviral medications within the last 30 days.
* Chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent >= 10 mg/day).
* Known hypersensitivity to sofosbuvir and velpatasvir, or formulation excipients.
* Hepatocellular carcinoma, or the presence of a mass on imaging studies of the liver that is suggestive of hepatocellular carcinoma, or an alpha-fetoprotein level of greater than 500 mg/mL
* Active psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, or personality disorder that, in the investigator s opinion, might interfere with participation in the study.
* Presence of conditions that, in the opinion of the investigators, would not allow the subject to n the current study for at least 1 year.

Phase II Follow-up

* Pregnancy
* Current or prior history of any of the following:

  * Clinically significant illness (other than resolved HCV) or any other major medical disorder that may interfere with subject treatment, assessment, or compliance with the protocol; subjects currently under evaluation for a potentially clinically significant illness

(other than HCV) are also excluded

--Decompensated liver disease as defined by serum bilirubin >= 2.5 mg/dL (with direct

bilirubin >= 1.5 mg/dL), INR >1.5 a serum albumin of less than 3 g/dL, or a history of ascites, hepatorenal syndrome, variceal bleeding, or hepatic encephalopathy.

* Solid organ transplantation
* Significant pulmonary disease, significant cardiac disease

  * History of malignancy or treatment for a malignancy within the past 3 years that is associated with a life expectancy <5 years (except adequately treated carcinoma in situ or basal cell carcinoma of the skin)
  * Chronic liver disease with the exception of steatosis (e.g., chronic hepatitis B, hemochromatosis, Wilson s disease, alfa-1 antitrypsin deficiency, cholangitis)
  * Evidence of harmful or hazardous drinking as defined as a score >= 8 on the AUDIT questionnaire
  * Co-infection with HIV defined as the presence of anti-HIV in serum
  * Clinically relevant drug abuse based on patient history within 12 months of screening
  * Chronic use of systemically administered immunosuppressive agents (e.g., prednisone equivalent >= 10 mg/day)
  * Hepatocellular carcinoma, or the presence of a mass on imaging studies of the liver that is suggestive of hepatocellular carcinoma, or an alpha-fetoprotein level of greater than 500 mg/mL
  * Active psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, or personality disorder that, in the investigator s opinion, might interfere with participation in the study
  * Presence of conditions that, in the opinion of the investigators, would not allow the patient to be followed in the current study for at least 1 year.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase II: Liver-related clinical outcome, HCC, or liver-related mortality | 480 Weeks
  Composite of ascites, spontaneous bacterial peritonitis, hepatic encephalopathy, variceal hemorrhage, hepatocellular carcinoma, liver-related mortality
Phase I - SVR 12 | 24 weeks
  SVR at 12 weeks after completion of 12 weeks of treatment

SECONDARY OUTCOMES:
Phase II: All-cause mortality | 480 weeks
Phase II: Change in Fibroscan | 480 weeks
Phase II: Assess Regression in Portal Hypertension | 480 weeks
Phase II: HCC | 480 weeks
Phase II: Change in Ishak fibrosis score | 480 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-DK-0091.html